CLINICAL TRIAL: NCT04408677
Title: Normative Data Collection Study of the Zilia Ocular for the Measurement of Oxygen Saturation in the Retina
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator and Sponsor expectations for the study not aligned, along with time conflicts for study completion. Discontinuation of the study is not related to the safety and/or effectiveness of the device.
Sponsor: Zilia Inc. (Industry)
Collaborators: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZCI01
Record Dates: First submitted 2020-05-15; First posted 2020-05-29 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Retinal Vascular; Retina

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Normative data (Experimental): Ocular oxygen saturation non-invasively measured at 3 eye fundus locations in the participant's right eye
  Interventions: Device: Zilia Ocular
- Repeatability (Experimental): Ocular oxygen saturation non-invasively measured at 3 eye fundus locations in the participant's right eye. After a 15 to 30 minutes break, same measurements repeated.
  Interventions: Device: Zilia Ocular
- Inter-eye variability (Experimental): Ocular oxygen saturation non-invasively measured at 3 eye fundus locations in the participant's right eye. After a 15 to 30 minutes break, same measurements repeated in the left eye.
  Interventions: Device: Zilia Ocular

INTERVENTIONS:
Device: Zilia Ocular — Measurement of the oxygen saturation in the eye fundus

SUMMARY:
Mainstream oximetry devices use two-wavelength systems to photograph the retina and estimate the oxygen saturation levels in the retinal vessels by comparing light absorption in the blood of the vessels at the selected wavelengths. This method limits the measurements to large retinal vessels, depends heavily on calibration and is non-reproducible across machines. The few numbers of wavelengths used (two) also makes it very susceptible to noise (such as cataract). These shortcomings have largely limited the use of retinal oximetry in clinical practice.

A new technology for retinal oximetry has recently been developed to address issues of dual-wavelength oximeters. Zilia Ocular's oximetry machine uses multi-wavelengths of light to take continuous oxygenation measurements of any targeted regions of the retina. It can measure any area of the retina, including the blood vessels, retinal tissues and the optic nerve head. Its multi-wavelength design also allows it to be less susceptible to noise, more precise and reproducible. This technology has the potential to extend our understanding of retinal pathologies, serve as a new marker for retinal health and even be used as a diagnostic tool to detect retinal injuries before they become visible.

Zilia's novel technology is one of its kind, allowing continuous and accurate measurements of the retina's oxygen saturation. In order to apply this technology to study and investigate retinal diseases, we need to first examine its performance in normal eyes and build a normative database as a reference. Thus, the purpose of the current study is to build a database of baseline oximetry values in healthy Caucasian subjects. The reproducibility of the measurements will also be studied in a subset of patients.

DETAILED DESCRIPTION:
STUDY OBJECTIVES

Objectives

Primary:

1. To measure the oxygen saturation at different locations on the retina (macula, optic nerve head, nasal retina) in order to provide the range of these values in normal eyes.

Secondary:

1. To assess the repeatability of the device's measurements (on a subset of patients).
2. To assess the variability of measurements between the two eyes (on a subset of patients).

Outcomes

Primary Outcome:

1. Normative values of the retinal oxygen saturation at different locations on the retina.

Secondary Outcomes:

1. Intraclass correlation coefficient of the measurements on the same patient at the same visit.
2. Percent difference between the measurements of the two eyes.

STUDY HYPOTHESES

Primary:

1. Oxygen saturation should have a consistent range among healthy subjects.

Secondary:

1. Intraclass classification (ICC) between two measurements on the same eye of the same participant should be at least 90%.
2. Measurements between the two eyes should have a percent difference less than 5%.

STUDY DESIGN

Type of study: single-center.

Expected number of subjects:

For primary objective: N=120 subjects For secondary objective #1: n= 62 For secondary objective #2: n= 12

ELIGIBILITY:
Inclusion Criteria:

* Adult patients above 18 years old, able to consent and willing to undergo mydriasis.
* Caucasian descent.
* Intraocular pressure ≤ 21 mmHg.
* Normal ophthalmological exam.

Exclusion Criteria:

* Any history of systemic disease, which could affect the eye or oxygen levels (eg: diabetes, severe cardiovascular or respiratory disease).
* History of epilepsy.
* Prior intraocular surgery (except cataract surgery).
* Any history or signs of retinal or optic nerve diseases.
* Pregnancy, or breastfeeding.
* Familial history of glaucoma.
* Ametropia > 6 Diopters.
* Pupil dilation < 3.6 mm.
* Current smoker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-09-22 (Actual)

PRIMARY OUTCOMES:
Normative values of the retinal oxygen saturation at different locations on the retina | 12-15 months
  Oxygen saturation measurement in the eye fundus of healthy subjects from different age groups

SECONDARY OUTCOMES:
Intraclass correlation coefficient of the measurements on the same patient at the same visit | 12-15 months
  Repeatability of the eye fundus oxygen saturation measurements (same subject, same visit, same eye, same eye fundus location)
Percent difference between the measurements of the two eyes. | 12-15 months
  Variability of the eye fundus oxygen saturation measurements between the right and left eyes (same subject, same visit, different eye, same eye fundus location)

CONTACTS AND LOCATIONS:
Overall Officials: Béatrice Des Marchais, MD, Principal Investigator — CHU de Québec
Locations (1):
- Hôpital du Saint-Sacrement, Québec, Canada

IPD SHARING:
Plan to Share IPD: No